CLINICAL TRIAL: NCT02787876
Title: Efficacy and Safety of Pegteograstim on Chemotherapy-induced Neutropenia in Children With Solid Tumors
Brief Title: Pegteograstim in Children With Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-12-121
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2017-09

CONDITIONS: Chemotherapy Induced Neutropenia; Pediatric Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy induced neutropenia (Experimental): Pegteograstim 100 ug/kg (maximum 6 mg) on day 7 of the chemotherapy cycle
  Interventions: Drug: Pegteograstim

INTERVENTIONS:
Drug: Pegteograstim

SUMMARY:
To evaluate the efficacy and safety of pegteograstim on chemotherapy-induced neutropenia in children with solid tumors

DETAILED DESCRIPTION:
Children with solid tumor experience neutropenia after cytotoxic chemotherapy, and they usually receive granulocyte colony-stimulating factor (G-CSF) to stimulate neutrophil recovery. However it needs daily injection of G-CSF. Pegteograstim is a new formulation of PEGylated recombinant human G-CSF analogue pegfilgrastim. In this study, investigators aimed to evaluate the efficacy and safety of pegteograstim on chemotherapy-induced neutropenia in children with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumor who undergo chemotherapy with carboplatin, etoposide, doxorubicin, cyclophosphamide (CEDC) and ifosfamide, carboplatin, etoposide (ICE) regimen

Exclusion Criteria:

* Patients with organ dysfunction (creatinine > 2mg/dL, ejection fraction <40% or severe arrhythmia/conduction disorder, other severe organ dysfunction)
* Hypersensitivity to pegteograstim, protein originated from E-coli, pegfilgrastim, filgrastim or latex.
* Patients with bleeding tendency to whom subcutaneous injection should be avoided.
* Active infection or infectious fever during the screening period.
* Genetic problem to fructose tolerance.
* Patients who participated in other clinical trial within 4 weeks before enrollment.
* Pregnant and nursing women

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-10-04 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events | Up to 3 weeks after the injection of pegteograsim
Duration of neutropenia (absolute neutrophil count (ANC) < 500/uL) | Up to 6 weeks

SECONDARY OUTCOMES:
Duration of severe neutropenia (ANC < 100/uL) | Up to 6 weeks
Lowest value of ANC | Up to 6 weeks
Days with neutropenic fever | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Cho HW, Lee JW, Ju HY, Hyun JK, Yoo KH, Koo HH, Kim K, Sung KW. Safety and Efficacy of Pegteograstim on Chemotherapy-induced Neutropenia in Children and Adolescents With Solid Tumors. J Pediatr Hematol Oncol. 2022 Mar 1;44(2):e362-e367. doi: 10.1097/MPH.0000000000002206. PMID 34010932